CLINICAL TRIAL: NCT04723797
Title: The Effect of a Physical Activity Program on Burnout Risk Among Secondary School: a Randomised Controlled Trial
Brief Title: The Effect of a Physical Activity Program on Burnout Risk Among Secondary School Teachers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Luna Coffyn, Master student, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B.U.N. 1432020000307
Record Dates: First submitted 2021-01-15; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Burnout Risk; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized control trial with a control group, a moderate-intensity intervention group, and a high-intensity intervention group
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): The participants in the control group will be asked to maintain their lifestyle as before the study.
- Moderate-intensity group (Experimental): Participants will be asked to perform a physical activity program, consisting of cycling and/or running for 6 weeks of at least 150min/week. This at a moderate intensity, which means a slightly increased heart rate and breathing also talking is possible.
  Interventions: Other: Physical activity
- Vigorous-intensity group (Experimental): Participants will be asked to perform a physical activity program, consisting of cycling and/or running for 6 weeks of at least 75min/week. This at a vigorous intensity, which means increased heart rate and breathing also talking is possible.
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — Physical activity program consisting of running and/or cycling
  Arms: Moderate-intensity group; Vigorous-intensity group

SUMMARY:
The purpose of this study is to assess the effect of a 6 weeks physical activity program on burnout risk in secondary school teachers. Also, the difference between the effects of moderate en vigorous-intensity physical activity will be investigated.

DETAILED DESCRIPTION:
Given the increased risk of burnout among secondary school teachers, effective interventions are needed. Physical activity may play a big role in preventing and/or reducing burnout. Therefore the purpose of this research is to investigate the effect of physical activity on the risk of burnout in secondary school teachers. The participants in the intervention group will be asked to perform a specific physical activity program (including running and/or cycling at a moderate or vigorous intensity) for 6 weeks. The control group will be asked to keep their lifestyle as it was prior to the study. To assess the effect of this activity program, the participants will have to fill in a questionnaire at three time points. Lastly, the participants have to fill in an activity diary every day, enabling to assess intervention adherence.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are not meeting the guidelines for physical activity.
* Participants who are willing to run or cycle.

Exclusion Criteria:

* Participants who are not speaking the Dutch language.
* Participants unable or unwilling to give informed consent.
* Participants who are not able to be physically active, due to injuries, physical disabilities, etc.
* Participants who already met the guidelines for physical activity.
* Participants who are following a diet.
* Participants who have been following psychological treatment in the past 6 months.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-04-04 (Estimated); Study Completion 2021-04-25 (Estimated)

PRIMARY OUTCOMES:
Burnout risk | 9 weeks
  Assessing the burnout risk by using the Burnout assessment tool (BAT). It consist 34 items scored on a 5-Point likert scale ranging from 1 (never) to 5 always. The greater the total score, the more the participant is in risk of a burnout.
Recovery need | 9 weeks
  Assessing the recovery need by using the Short Inventory to Monitor Psychosocial. hazards (SIMPH). This survey consists of 5 questions with the answer options 'yes' or no'. A score of 3 times 'yes' out of 5, is an indication of a possible increased need for recovery at work.

SECONDARY OUTCOMES:
School and teaching subjects | 9 weeks
  It is a self-designed questionnaire about location and type of school, grades and teaching subjects
Rate of perceived exertion | 9 weeks
  Effort and exertion will be measured by using the Borg Rating of Perceived Exertion scale. The borg scale ranges from '6' to '20' and is highly correlated with the heart rate. A borg scale of 10 corresponds to a heart rate of 100bpm in a healthy adult.

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided